CLINICAL TRIAL: NCT06185179
Title: Use of Metformin to Improve Muscle Regrowth in Older Adults
Brief Title: Metformin and Muscle Recovery
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Micah Drummond, Professor, Physical Therapy and Athletic Training, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 086328
Record Dates: First submitted 2023-12-13; First posted 2023-12-29 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Muscle Atrophy or Weakness
MeSH Terms: conditions — Muscular Atrophy; Asthenia | interventions — Metformin

STUDY DESIGN:
Intervention Model Description: 2-weeks single leg immobilization followed by 2-weeks of recovery
Who Masked: Participant, Investigator
Masking Description: Metformin and Placebo pills will be encapsulated by the pharmacy in order to protect treatment assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Metformin (Experimental): Metformin pills will be given orally and daily during the 2-week recovery period following single leg immobilization Metformin will be titrated up to a dose 2g/day. 1g dose (two 500 mg pills) will be taken in the morning and a 1g dose will be taken in the evening. This will take place over each day for 14 days during the recovery period.
  Interventions: Drug: Metformin
- Placebo (Placebo Comparator): Placebo pills will be given orally and daily during the 2-week recovery period following single leg immobilization. Two pills will be taken in the morning and two pills will be taken in the evening. This will take place over each day for 14 days during the recovery period.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Metformin — Metformin will be distributed in 500mg pills.
  Other Names: Glucophage; Fortamet; Glumetza; Riomet
  Arms: Metformin
Other: Placebo — Placebo will be distributed in pill form
  Arms: Placebo

SUMMARY:
A hallmark of aging is an impaired ability to adequately recover following a stressor, such as muscle disuse, resulting in muscle fibrosis and weakness thereby increasing the risk for falls and loss of independence. Mechanistic-based therapeutic strategies to enhance muscle recovery in older adults do not exist. Metformin has been implicated to have positive effects on muscle size and function through non-glycemic mechanisms. Metformin has been shown to enhance macrophage function and lessen cellular senescence burden by targeting SASP in a variety of muscle interstitial cells. However, the role of metformin to improve muscle recovery in older adults following disuse atrophy through immunomodulating and senomorphic mechanisms have not been examined. Therefore, the purpose of this study is to conduct a randomized, double blind, placebo-controlled clinical trial in older adult participants to determine if short-term metformin delivery (vs placebo) during the recovery phase following disuse atrophy can improve muscle regrowth.

DETAILED DESCRIPTION:
Aging is associated with impaired muscle recovery following disuse atrophy. If not addressed, restricted muscle regrowth and function may lead to a cascade of health crisis events for the aged individual (falls, disability, metabolic diseases). Clinically adopted treatments that promote muscle recovery, particularly in elderly patients, do not exist. The long-term goal of this project is to develop mechanistic-based therapeutic approaches to accelerate muscle recovery following disuse atrophy in older adults.

Macrophages are well understood to play a requisite role in myofiber remodeling including removal of debris and senescent cells, promotion of stem/satellite cell proliferation and differentiation, and regulation fibro-adipogenic progenitor cell (FAP) dynamics and fate. It is known that aged muscle during recovery have an impaired macrophage inflammatory and functional response complimented with poor muscle recovery. The investigators posit that age-related local immune dysfunction disrupts extracellular matrix (ECM) remodeling following muscle disuse by reducing the removal of senescence cells resulting in their accumulation. Therefore, treatments are needed to improve macrophage function and mitigate cellular senescence to facilitate muscle cellular remodeling events (e.g., macrophage, satellite cells, FAPs) during recovery following disuse in aging.

Metformin has gained traction to be repurposed as a treatment for a broad range of age-related diseases but its role in regulating muscle regrowth following disuse atrophy in humans is not known. Metformin has shown to modulate inflammatory profiles, mitigate cellular senescence and SASP (e.g., macrophages, FAPs, and myoblasts) while also improving muscle regeneration and satellite cell function in injured mice. Therefore, metformin treatment could have therapeutic value to temper unwanted collagen deposition and promote muscle regrowth and function when strategically delivered during the muscle regrowth phase in aging by targeting immune cell function and cellular senescence and SASP.

The overarching hypothesis is that metformin would mitigate cellular senescence and SASP specifically in macrophages, FAPs and satellite cells and would correspond to enhanced muscle function following disuse atrophy. The investigators will conduct a randomized, placebo-controlled clinical trial in healthy older participants to test if metformin provided during a 14d recovery phase following unilateral limb immobilization would improve muscle macrophage, FAP and satellite cell function, reduce cellular senescence and muscle fibrosis.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 60y and older
2. BMI: <30 kg/m2
3. Good general medical health, ambulatory and in independent living setting
4. Adequate upper body strength to use assistive walking device (crutches, walker, etc) as assessed by PI/staff during screening
5. Clinical Frailty Scale score < 3
6. Mini-Cog score > 3

Exclusion Criteria:

1. History of cardiovascular disease (e.g., CHF, CAD, MI, CVA)
2. History of endocrine or metabolic disease such as hypo/hyperthyroidism and diabetes (Treated hypo/hyperthyroid for at least 6 months will be permitted)
3. History of kidney disease or failure (CKD > stage 4; serum creatinine >1.5mg/dL)
4. History of vascular disease
5. Risk of DVT including family history of thrombophilia, DVT, pulmonary emboli, myeloproliferative diseases including polycythemia (Hb>18 g/dL) or thrombocytosis (platelets>400x103/mL), and connective tissue diseases (positive lupus anticoagulant), hyperhomocystinemia, deficiencies of factor V Leiden, proteins S and C, and antithrombine III
6. Use of anticoagulant therapy (e.g., Coumadin, heparin)
7. Uncontrolled hypertension - Elevated systolic pressure >150 or a diastolic blood pressure > 100
8. Implanted electronic devices (e.g., pacemakers, electronic infusion pumps, stimulators)
9. Cancer or history of successfully treated cancer (less than 1 year) other than basal cell carcinoma
10. Chronic systemic corticosteroid use (≥ 2 weeks) within 4 weeks of enrollment and for study duration (intra-articular/topical/inhaled therapeutic or physiologic doses of corticosteroids will be permitted)
11. Androgens or growth hormone within 6 months of enrollment and for study duration (topical physiologic androgen replacement will be permitted)
12. Inability to abstain from smoking or vaping for duration of study
13. Currently taking estrogen products (topical estrogen products will be permitted)
14. Currently on weight loss diet or medication
15. History of stroke with motor disability
16. A recent history (<12 months) of GI bleed
17. History of liver disease or AST/ALT 2 times above the normal limit
18. History of respiratory disease (acute upper respiratory infection, history of chronic lung disease)
19. Any staff members who report directly to the principal investigators

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2029-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
% recovery of thigh muscle volume (TMV) | Thigh muscle volume will be determined at 14 days of single leg immobilization and at 14 days of recovery.
  recovery of thigh muscle volume will be defined as the percentage of TMV at recovery when comparing to the TMV immobilization time point ((TMV recovery - TMV immobilization)/TMV immobilization)*100.
  Thigh muscle volume will be determined by MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Micah Drummond, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No
IPD can be requested by the PI, Dr. Drummond.